CLINICAL TRIAL: NCT05286788
Title: Phase 2 Study of the MEK Inhibitor MEKTOVI® (Binimetinib) for the Treatment of Pediatric Adamantinomatous Craniopharyngioma
Brief Title: MEKTOVI® for the Treatment of Pediatric Adamantinomatous Craniopharyngioma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: Children's Hospital Colorado (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CONNECT2108
Record Dates: First submitted 2022-03-01; First posted 2022-03-18 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-03

CONDITIONS: Adamantinous Craniopharyngioma; Recurrent Adamantinomatous Craniopharyngioma
MeSH Terms: conditions — Craniopharyngioma | interventions — binimetinib

STUDY DESIGN:
Intervention Model Description: MEKTOVI® (binimetinib)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Stratum 1 and Stratum 2 (Experimental): Stratum 1: Patients with progressive or recurrent adamantinomatous craniopharyngiomas following radiation therapy.
  Stratum 2: Patients with measurable adamantinomatous craniopharyngioma who have undergone surgery but have not previously received radiation therapy. Progressive disease is allowed but not required
  Interventions: Drug: Binimetinib Oral Tablet [Mektovi]

INTERVENTIONS:
Drug: Binimetinib Oral Tablet [Mektovi] — Binimetinib oral continuous dosing 32 mg/m2 PO BID for 4 weeks
  Other Names: MEKTOVI

SUMMARY:
MEKTOVI (binimetinib) is an oral, highly selective reversible inhibitor of mitogen-activated extracellular signal regulated kinase 1 (MEK1) and MEK2. The biological activity of binimetinib that has been evaluated bith in vitro and in vivo in a wide variety of tumor types In this Phase II, the drug will be used to treat pediatric patients diagnosed with recurrent Adamantinomatous Craniopharyngioma including patients who have undergone surgery and/or radiation therapy.

DETAILED DESCRIPTION:
Adamantinomatous Craniopharyngioma (ACP) is a highly debilitating pediatric brain tumor that lacks medical anti-tumor therapies. Current therapy, which depends largely on surgery and radiation, is associated with poor quality of life and becomes more challenging and risky in the setting of recurrent disease. Recent discoveries regarding the biological characteristics of ACP indicate that available agents, including Mitogen-activated protein kinase/extracellular signal-regulated kinase (MAPK/ERK) pathway inhibitors may have efficacy in the control of ACP. Binimetinib is one such agent.

In this study, up to 38 patients will receive oral binimetinib at the recommended phase 2 pediatric dose (RP2D) of 32 mg/m2/dose PO every 12 hours for 4 weeks which represents one cycle. Cycles will last 28 days and treatment may continue for up to two years (26 cycles).

It will be a multi-center Phase 2 trial with two strata for patients aged >1 year and <25 years with measurable ACP who may have been previously treated with radiation (Stratum 1, 18 patients) or without radiation (Stratum 2, 18 patients).

ELIGIBILITY:
Inclusion Criteria:

1. Age: Patients must be ≥ 12 months and ≤ 39 years of age at the time of study enrollment.
2. Diagnosis: Patients with histologically-confirmed adamantinomatous craniopharyngioma (ACP) Histologic confirmation of ACP may be made on solid tumor or, if no solid tumor can be safely obtained, cyst fluid with classic ACP characteristics of thick, cholesterol-rich, greenish-brown liquid in the context of imaging features consistent with craniopharyngioma, including lobulated, cystic/solid mass with calcifications that originates in the sellar/suprasellar region.
3. Disease Status: Patients must have measurable disease.

   * Stratum 1: Patients with progressive or recurrent ACP who demonstrate cystic and/or solid recurrence or progression at least 6 months post completion of radiation therapy
   * Stratum 2: Patients with measurable ACP who have undergone surgery but have NOT previously undergone irradiation (but may have received prior systemic or intracystic therapy). Progressive disease is allowed but not required.
4. Performance Level: Karnofsky ≥ 50% for patients > 16 years of age and Lansky ≥ 50 for patients ≤ 16 years of age (See Appendix I). Note: Neurologic deficits in patients with CNS tumors must have been stable for at least 7 days prior to study enrollment. Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
5. Prior Therapy: Patients must have recovered or stabilized from the acute toxic effects of prior treatments

   * Biologic (anti-neoplastic agent): At least 7 days must have elapsed after the last (systemic or intracystic) dose of a biologic agent. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur. The duration of this interval must be discussed with the study chair
   * Immunotherapy: At least 42 days after the completion of any type of systemic immunotherapy, e.g. tumor vaccines.
   * Monoclonal antibodies: At least 21 days after the last dose of a monoclonal antibody.
   * Radiation therapy: Patients must have had their last (conventional or hypofractionated) fraction of: a) Focal irradiation > 6 months prior to enrollment and b) No prior craniospinal irradiation is permitted.
   * Corticosteroids: Patients receiving dexamethasone must be on a stable or decreasing dose for at least 1 week prior to enrollment
   * Myelosuppressive systemic therapy: At least 21 days must have elapsed after the last systemic myelosuppressive therapy.
   * Surgery: At least 6 weeks must have elapsed since major or intermediate surgery. Major surgery includes major craniotomy for tumor resection of cyst fenestration, organ resection, and exploratory laparotomy. Intermediate procedures include ventriculoperitoneal shunt placement, stereotactic brain biopsy, and intraventricular catheter placement. Minor procedures that are not excluded include skin biopsy/incision and drainage, bone marrow aspirate, and central venous catheter placement, ommaya aspirations, lumbar punctures, and nasal endoscopy to remove packing.
6. Organ Function Requirements

   Adequate Bone Marrow Function Defined as:
   * Peripheral absolute neutrophil count (ANC) ≥1000/mm3
   * Platelet count ≥100,000/mm3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment)
   * Hemoglobin >8 g/dL (may be transfused)

   Adequate Renal Function Defined as:
   * Creatinine clearance or radioisotope GFR > 70ml/min/1.73 m2 or
   * A serum creatinine based on (Schwartz et al. J. Peds, 106:522, 1985) age/gender as follows:

     1. to < 2 years: maximum serum creatinine 0.6 mg/dL for males and females. 2 to < 6 years: maximum serum creatinine 0.8 mg/dL for males and females. 6 to < 10 years: maximum serum creatinine 1.0 mg/dL for males and females. 10 to < 13 years: maximum serum creatinine 1.2 mg/dL for males and females. 13 to < 16 years: maximum serum creatinine 1.5 mg/dL for males and 1.4 mg/dL for females. ≥ 16 years: maximum serum creatinine 1.7 mg/dL for males and 1.4 mg/dL for females.

   Adequate Liver Function Defined as:
   * Total bilirubin ≤ 1.5 × institutional upper limit of normal
   * AST (SGOT) ≤ 2.5 × institutional upper limit of normal
   * ALT (SGPT) ≤ 2.5 × institutional upper limit of normal

   Adequate Cardiac Function Defined as:
   * Left Ventricular Ejection Fraction greater than the institutional lower limit of normal by echocardiogram
   * QTc ≤ 480 msec (by Bazett formula)

   Adequate Neurologic Function Defined as:
   * Patients with neurological deficits should have deficits that are stable for a minimum of 1 week prior to enrollment.
   * Patients with current seizure disorders may be enrolled if seizures are well-controlled on antiepileptic therapies.
7. Informed Consent: All patients and/or their parents or legally authorized representatives must sign a written informed consent. Assent, when appropriate, will be obtained according to institutional guidelines

Exclusion Criteria:

1. Pregnancy or Breast-Feeding: Pregnant or breast-feeding women will not be entered on this study due to unknown risks of fetal and teratogenic adverse events as seen in animal/human studies. Pregnancy tests must be obtained in girls who are post-menarchal. Males or females of reproductive potential may not participate unless they have agreed to use an effective contraceptive method for at least 90 days after discontinuation of drug for females and at least 60 days for males. For females of childbearing potential, agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods (bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices; hormonal contraceptive methods must be supplemented by a barrier method) and agreement to refrain from donating eggs are required. For males of reproductive potential, agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agreement to refrain from donating sperm.
2. Gastrointestinal Disease:

   * Patients with a history of serious gastrointestinal disease, including inflammatory bowel disease or gastrointestinal perforation
   * Patients who are unable to absorb enteral medications
   * Administration via NG/NJ/G-tube is allowed
3. Concomitant Medications

   * Corticosteroids: Patients receiving corticosteroids who have not been on a stable or decreasing dose of corticosteroid for at least 7 days prior to enrollment are not eligible.
   * Investigational Drugs: Patients who are currently receiving another investigational drug are not eligible.
   * Anti-cancer Agents: Patients who are currently receiving other anti-cancer agents are not eligible.
4. Study Specific:

   * Patients who have an uncontrolled infection are not eligible.
   * Patients who have received any live or attenuated vaccinations within three months prior to start of therapy are not eligible.
   * Any significant concurrent medical or surgical condition that would jeopardize the patient's safety or ability to complete the study, including, but not limited to, disease of the nervous, renal, hepatic, cardiac (such as symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia), pulmonary, or endocrine system
   * Patients who have a history of Human Immunodeficiency Virus, Hepatitis B Virus, Hepatitis C Virus or Tuberculosis infection are not eligible.
   * Patients who have received a prior solid organ transplantation are not eligible.
   * Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible.
   * Patients who have a history of alcohol, drug, or chemical abuse within 6 months of screening.
   * Patients who have had surgery within the last 6 weeks or who have concerns for poor postsurgical wound healing.
   * Patients who have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to tocilizumab and its excipients are not eligible.

Ages: 1 Year to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-04-10 (Actual); Primary Completion 2027-04-10 (Estimated); Study Completion 2027-04-10 (Estimated)

PRIMARY OUTCOMES:
Sustained objective response rate of patients with recurrent/progressive previously irradiated ACP to treatment with oral binimetinib | From Day 1 of treatment through 30 days following end of protocol treatment
  To calculate the number of patients who experience sustained objective response rate [minor response (MR) + partial response (PR) + complete response (CR)] of patients with recurrent/progressive previously irradiated Adamantinomatous Craniopharyngioma to treatment with oral binimetinib (Stratum 1).
Sustained objective response rate of patients with measurable ACP who have undergone surgery but have not been previously treated with radiation to treatment with oral binimetinib | From Day 1 of treatment through 30 days following end of protocol treatment
  To calculate the number of patients who experience sustained objective response rate (MR + PR + CR) of patients with measurable Adamantinomatous Craniopharyngioma who have undergone surgery but have not been previously treated with radiation to treatment with oral binimetinib (Stratum 2).

SECONDARY OUTCOMES:
Biological effects of binimetinib on ACP tumor tissue and cyst fluid. | From Day 1 of treatment through 30 days following end of protocol treatment
  To measure concentrations of various chemokines including IL-6, IL-8, IL-10 and CXCL1in cyst fluid or tumor or blood of ACP patients treated with binimetinib. Comparisons will be made with known levels in the literature and among patient samples from within the study.
Toxicities associated with tocilizumab in children with ACP | 24 months
  To calculate the number of participants with, as well as frequency and severity of, binimetinib-related Adverse Events as assessed by CTCAE v5.0 in children with recurrent or refractory ACP
PFS of ACP patients treated with binimetinib after radiation | 12 months
  To assess one-year progression-free survival (PFS) rates for patients with ACP who are treated with binimetinib following progression after radiation (Stratum 1).
PFS of ACP patients treated with binimetinib who have not received radiation | 12 months
  To assess one-year progression-free survival (PFS) rates for patients with ACP who are treated with binimetinib who have not previously received radiation (Stratum 2).

CONTACTS AND LOCATIONS:
Overall Officials: Holly Lindsay, MD, Study Chair — Children's Hospital Colorado; Todd C Hankinson, MD, Study Chair — Children's Hospital Colorado; Maryam Fouladi, MD, Principal Investigator — Nationwide Children's Hospital
Locations (10):
- United States (5):
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Nicklaus Children's Hospital, Miami, Florida
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
- Australia (3):
  - Sydney Children's Hospital, Randwick, New South Wales
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Perth Children's Hospital, Perth, Western Australia
- Canada (2):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CHU Sainte-Justine, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Foreman NK, Faestel PM, Pearson J, Disabato J, Poole M, Wilkening G, Arenson EB, Greffe B, Thorne R. Health status in 52 long-term survivors of pediatric brain tumors. J Neurooncol. 1999 Jan;41(1):47-53. doi: 10.1023/a:1006145724500. PMID 10222422
- [Background] Goldman S, Pollack IF, Jakacki RI, Billups CA, Poussaint TY, Adesina AM, Panigrahy A, Parsons DW, Broniscer A, Robinson GW, Robison NJ, Partap S, Kilburn LB, Onar-Thomas A, Dunkel IJ, Fouladi M. Phase II study of peginterferon alpha-2b for patients with unresectable or recurrent craniopharyngiomas: a Pediatric Brain Tumor Consortium report. Neuro Oncol. 2020 Nov 26;22(11):1696-1704. doi: 10.1093/neuonc/noaa119. PMID 32393959
- [Background] Apps JR, Carreno G, Gonzalez-Meljem JM, Haston S, Guiho R, Cooper JE, Manshaei S, Jani N, Holsken A, Pettorini B, Beynon RJ, Simpson DM, Fraser HC, Hong Y, Hallang S, Stone TJ, Virasami A, Donson AM, Jones D, Aquilina K, Spoudeas H, Joshi AR, Grundy R, Storer LCD, Korbonits M, Hilton DA, Tossell K, Thavaraj S, Ungless MA, Gil J, Buslei R, Hankinson T, Hargrave D, Goding C, Andoniadou CL, Brogan P, Jacques TS, Williams HJ, Martinez-Barbera JP. Tumour compartment transcriptomics demonstrates the activation of inflammatory and odontogenic programmes in human adamantinomatous craniopharyngioma and identifies the MAPK/ERK pathway as a novel therapeutic target. Acta Neuropathol. 2018 May;135(5):757-777. doi: 10.1007/s00401-018-1830-2. Epub 2018 Mar 14. PMID 29541918
- [Background] Haston S, Pozzi S, Carreno G, Manshaei S, Panousopoulos L, Gonzalez-Meljem JM, Apps JR, Virasami A, Thavaraj S, Gutteridge A, Forshew T, Marais R, Brandner S, Jacques TS, Andoniadou CL, Martinez-Barbera JP. MAPK pathway control of stem cell proliferation and differentiation in the embryonic pituitary provides insights into the pathogenesis of papillary craniopharyngioma. Development. 2017 Jun 15;144(12):2141-2152. doi: 10.1242/dev.150490. Epub 2017 May 15. PMID 28506993
- [Background] Bendell JC, Javle M, Bekaii-Saab TS, Finn RS, Wainberg ZA, Laheru DA, Weekes CD, Tan BR, Khan GN, Zalupski MM, Infante JR, Jones S, Papadopoulos KP, Tolcher AW, Chavira RE, Christy-Bittel JL, Barrett E, Patnaik A. A phase 1 dose-escalation and expansion study of binimetinib (MEK162), a potent and selective oral MEK1/2 inhibitor. Br J Cancer. 2017 Feb 28;116(5):575-583. doi: 10.1038/bjc.2017.10. Epub 2017 Feb 2. PMID 28152546
- [Background] Watanabe K, Otsu S, Hirashima Y, Morinaga R, Nishikawa K, Hisamatsu Y, Shimokata T, Inada-Inoue M, Shibata T, Takeuchi H, Watanabe T, Tokushige K, Maacke H, Shiaro K, Ando Y. A phase I study of binimetinib (MEK162) in Japanese patients with advanced solid tumors. Cancer Chemother Pharmacol. 2016 Jun;77(6):1157-64. doi: 10.1007/s00280-016-3019-5. Epub 2016 Apr 12. PMID 27071922
- [Background] Patel K, Allen J, Zagzag D, Wisoff J, Radmanesh A, Gindin T, Nicolaides T. Radiologic response to MEK inhibition in a patient with a WNT-activated craniopharyngioma. Pediatr Blood Cancer. 2021 Mar;68(3):e28753. doi: 10.1002/pbc.28753. Epub 2020 Oct 19. No abstract available. PMID 33073916
- See also: Mektovi prescribing information — http://labeling.pfizer.com/ShowLabeling.aspx?id=12988.
- See also: Mektovi product characteristics — https://www.ema.europa.eu/en/documents/product-information/mektovi-epar-product-information_en.pdf